CLINICAL TRIAL: NCT05311813
Title: Evaluation of Safety and Efficacy of Monotherapy Versus Polytherapy of Enoxaparin and Hydroxychloroquine for the Treatment of Covid-19
Brief Title: Safety and Efficacy of Enoxaparin and Hydroxychloroquine in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Raghda R.S. Hussein, Assistant Professor of Clinical Pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-21013
Record Dates: First submitted 2022-04-04; First posted 2022-04-05 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 infection; Enoxaparin; Hydroxychloroquine; ICU stay
MeSH Terms: conditions — COVID-19 | interventions — Enoxaparin; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Study Patients were randomized into four parallel equal groups using a computerized random number generator using simple randomization with an equal allocation ratio. Two hundred and twenty patients were eligible. Twenty patients were excluded due to not meeting the inclusion criteria (n=14) or the decline to be enrolled in the study (n=4). The sample size was calculated by G.power version 3.1 for windows (Faul et al., 2009). With a priori calculating the sample size based on the length of stay among the studied groups using one way ANOVA test (F-test group), at an effect size (0.306), alpha probability (0.05) and power (95%), the calculated sample size was 184 in the 4 groups that increased to 200 (with 6% increase) to overcome the missing of data and dropout or loss of follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): The control group including 50 patients (n=50) receiving the conventional therapy of Covid-19 adopted by the Egyptian ministry of health for 15 days.
  Interventions: Drug: Enoxaparin, Hydroxychloroquine
- Enaxoprin group (Active Comparator): The enoxaparin group (n=50) which received 40mg/day SC for 14 days (for patients with normal renal function and body weight between 50 and 100kg) plus the conventional therapy of Covid-19 adopted by the Egyptian ministry of health for 15 days.
  Interventions: Drug: Enoxaparin, Hydroxychloroquine
- Hydroxychloroquine group (Active Comparator): The HCQ group which received 400 mg/day HCQ for five days plus the conventional therapy of Covid-19 adopted by the Egyptian ministry of health for 15 days(n=50).
  Interventions: Drug: Enoxaparin, Hydroxychloroquine
- Enoxaparin plus Hydroxychloroquine group (Active Comparator): The HCQ plus Enoxaparin combination group including 50 patients receiving combined therapy of 400 mg/day HCQ for five days and 40mg/day enoxaparin for 14 days plus the conventional therapy of COVID-19 adopted by the Egyptian ministry of health for 15 days
  Interventions: Drug: Enoxaparin, Hydroxychloroquine

INTERVENTIONS:
Drug: Enoxaparin, Hydroxychloroquine — To compare efficiency and safety of Enoxaparin and Hydroxychloroquine as monotherapy versus Polytherapy

SUMMARY:
In this randomized controlled study, two hundred patients with positive PCR and laboratory confirmed COVID-19 will be classified randomly into four groups. The first group is the control group and will be given the conventional treatment of covid-19 only. The second group will be given enoxaparin plus the conventional treatment of Covid-19. The third group will be given hydroxychloroquine (HCQ 400 mg/day) for five days plus the conventional treatment of covid-19. The last group will be given combined therapy of HCQ 400 mg/day and enoxaparin plus the conventional therapy of covid-19

The efficacy will be assessed by the time of undetectable viral RNA, duration of treatment and length of hospital stay. The safety will be assessed by measuring the severity of side effects by following up the patients after treatment.

DETAILED DESCRIPTION:
Although numerous therapeutic agents for COVID-19 are under investigation, an effective therapy remains a challenge among researchers. To date, hydroxychloroquine has been widely used for covid-19 treatment, despite that its efficacy and safety need further investigations. Coagulopathies are major complications of covid-19 infection, hence prophylactic anticoagulation has been recommended in all hospitalized patients. This study aims to assess the efficacy and safety of Enoxaparin and hydroxychloroquine used separately or combined and added to standard care versus standard care alone in Covid-19 infected patients. An observational study including two hundred patients (98 males, 102 females) with laboratory confirmed covid-19 infection was conducted. Patients admitted to hospital were randomly allocated into four equal treatment groups. The first group received standard Covid-19 therapy, second group received enoxaparin 40mg/day SC for 14 days plus standard Covid-19 therapy, third group received 400 mg/day HCQ for five days plus standard Covid-19 therapy. The fourth group received a combination of 400 mg/day HCQ and enoxaparin plus standard Covid-19 therapy. The clinical disease course progression was evaluated by duration to a negative PCR, length of hospital or ICU stay, and mortality rate. The safety of treatments was evaluated by measuring liver biochemistries (ALT, AST), random blood glucose levels and adverse effects during the 28 days of treatment. Patients on Enoxaparin plus standard Covid-19 therapy significantly showed a decrease in length of hospital stay, ICU admission and mortality compared to all other treatments. However, the duration to both negative PCR and clinical improvement did not find any significance. These findings suggest that enoxaparin treatment was safe, effective, and well tolerated and has a role in decreasing the progression of the disease and its complications while HCQ did not discover any evidence of extra therapeutic benefits over other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed COVID-19 infection by PCR test within 7 days prior to admission or during admission to hospital, CT or radiographic findings of pneumonia. Clinically suspected infection by symptoms like loss of smell and taste. No medical history that may interfere with treatment or with this clinical trial.

Exclusion Criteria:

* Patient who had allergy or contraindication to HCQ, pregnant and lactating females, and patients with immune diseases, cardiac problem, had history of acute kidney injury or who received multiple cycles of anticoagulants were excluded from the study. Written informed consent was obtained from each participant. All study risks and benefits were thoroughly explained to patients' prior participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy | 6 monthes
  The hospital stay of COVID-19 patients

SECONDARY OUTCOMES:
Assessment of Safety | 6 monthes
  Mortality of COVID-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University teaching Hospital, Banī Suwayf, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP